CLINICAL TRIAL: NCT01412177
Title: A Prospective, Randomized, Double-blind, Placebo-controlled, Multicenter, Phase 2b Study of OTO-104 Given as a Single Intratympanic Injection in Subjects With Unilateral Meniere's Disease
Brief Title: OTO-104 for the Treatment of Meniere's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otonomy, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 104-201102
Record Dates: First submitted 2011-07-31; First posted 2011-08-09 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-08

CONDITIONS: Meniere's Disease
Keywords: Meniere's Disease; Vertigo; Definitive vertigo; Vertigo episodes; Vertigo frequency; Tinnitus; Hearing loss; Aural fullness
MeSH Terms: conditions — Meniere Disease; Vertigo; Tinnitus; Hearing Loss

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OTO-104 (Experimental)
  Interventions: Drug: OTO-104
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OTO-104 — Single intratympanic injection of 12 mg OTO-104
  Arms: OTO-104
Drug: Placebo — Single intratympanic injection of placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness of OTO-104 for the treatment of Meniere's disease.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of unilateral Meniere's disease by 1995 American Academy of Otolaryngology - Head and Neck Surgery (AAOHNS) criteria and reports active vertigo for the 2 months prior to the study lead-in period.
* Subject has experienced active vertigo during the lead-in period.
* Subject has documented asymmetric sensorineural hearing loss.
* Subject agrees to maintain their current treatments for Meniere's disease while on-study.
* Subjects currently on a low-salt diet and/or diuretic at the time of screening agree to continue this treatment throughout the study.

Exclusion Criteria:

* Subject is pregnant or lactating.
* Subject has a history of immunodeficiency disease.
* Subject has a history of previous endolymphatic sac surgery.
* Subject has a history of previous use of intratympanic (IT) gentamicin in the affected ear.
* Subject has a history of tympanostomy tubes with evidence of perforation or lack of closure.
* Subject has experienced an adverse reaction to IT injection of steroids.
* Subject has used an investigational drug or device in the 3 months prior to screening.
* Subject has previously been randomized to a trial of OTO-104.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2013-11; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Reduction in vertigo frequency as measure of efficacy of OTO-104 in subjects with Meniere's disease | 4 months

SECONDARY OUTCOMES:
Evaluation of adverse events, otoscopic exams, audiometry, Word Recognition Score and tympanometry as a measure of safety and tolerability | 4 months
Evaluation of tinnitus patient reported questionnaire and daily diary as a measure of impact of tinnitus on activities of daily living | 4 months
Evaluation of patient reported questionnaires as a measure of impact on patient daily activities | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Carl LeBel, PhD, Study Chair — Otonomy, Inc.
Locations (2):
- United States (2):
  - Many sites in US and Canada. Refer to the contact info listed below., San Diego, California
  - UC Health Otolaryngology - Head and Neck Surgery, Cincinnati, Ohio

REFERENCES:
- See also: Please click on this link for more information regarding this study and referral to the closest study site if you qualify (http://menieresresearchstudy.com). — http://menieresresearchstudy.com